CLINICAL TRIAL: NCT02123017
Title: An Observer-blinded, Dose-finding Study to Investigate the Safety, Efficacy, and Patient Preference of Lactulose for Oral Solution With Bisacodyl for Cleansing of the Colon as a Preparation for Colonoscopy in Adults
Brief Title: Efficacy and Safety of Bisacodyl and Lactulose as a Preparation for Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CPI-KR-005
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Colonoscopy Preparation
Keywords: Bowel Evacuation; Colonoscopy Preparation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 90 grams of Crystalline Lactulose (Experimental): 15 mg of bisacodyl, plus 30 grams of crystalline lactulose x three doses
  Interventions: Drug: 90 grams of Crystalline Lactulose
- 135 grams of Crystalline Lactulose (Experimental): 15 mg of bisacodyl, plus 45 grams of crystalline lactulose x three doses
  Interventions: Drug: 135 grams of Crystalline Lactulose
- 180 grams of Crystalline Lactulose (Experimental): 15 mg of bisacodyl, plus 60 grams of crystalline lactulose x three doses
  Interventions: Drug: 180 grams of Crystalline Lactulose

INTERVENTIONS:
Drug: 90 grams of Crystalline Lactulose — 15 mg of bisacodyl, plus 30 grams crystalline lactulose x 3 doses
  Arms: 90 grams of Crystalline Lactulose
Drug: 135 grams of Crystalline Lactulose — 15 mg of bisacodyl, plus 45 grams crystalline lactulose x 3 doses
  Arms: 135 grams of Crystalline Lactulose
Drug: 180 grams of Crystalline Lactulose — 15 mg of bisacodyl, plus 60 grams crystalline lactulose x 3 doses
  Arms: 180 grams of Crystalline Lactulose

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of bisacodyl combined with escalating doses of lactulose to be used as a preparation for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring bowel evacuation for colonoscopy.

Exclusion Criteria:

* Patients with galactosemia (galactose-sensitive diet).
* Patients known to be hypersensitive to any of the components of lactulose for oral solution.
* Patients with a known abnormality on screening or a vital sign assessments that, in the Investigator's judgment, may pose a significant risk including those pertaining to dehydration or electrolyte shifts.
* Patients with a history of impaired renal function.
* Patients with current or recent history of hypotension, as defined by the Investigator.
* Patients with a history of long Q-T syndrome.
* Patients with a history of a failed bowel preparation.
* Patients with severe constipation, defined as those patients taking daily prescription or over-the-counter laxatives.
* Patients with possible bowel obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon, ileus or previous colonic surgery (except hemorrhoidectomy and polypectomy).
* Patients on lactulose therapy or receiving any treatment for chronic constipation.
* Be pregnant or nursing.
* Patients expected to require electrocautery or argon plasma coagulation.
* Patients less than 18 years of age.
* Inability to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]) and agree to abide by the study restrictions.
* Be otherwise unsuitable for the study, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Krause, MD, Principal Investigator — ClinSearch, LLC
Locations (1):
- ClinSearch, LLC, Chattanooga, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 90 Grams Crystalline Lactulose: 15 mg bisacodyl, plus 30 grams crystalline lactulose x 3 doses
- 135 Grams Crystalline Lactulose: 15 mg bisacodyl, plus 45 grams crystalline lactulose x 3 doses
- 180 Grams Crystalline Lactulose: 15 mg bisacodyl, plus 60 grams crystalline lactulose x 3 doses
Period: Overall Study
Arm/Group | 90 Grams Crystalline Lactulose | 135 Grams Crystalline Lactulose | 180 Grams Crystalline Lactulose
Started | 8 | 12 | 12
Completed | 8 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients adhered to the one set of study-level eligibility criteria.
Groups:
- 90 Grams of Crystalline Lactulose: 15 mg of bisacodyl and 30 grams crystalline lactulose x 3 doses
- 135 Grams of Crystalline Lactulose: 15 mg of bisacodyl and 45 grams crystalline lactulose x 3 doses
- 180 Grams of Crystalline Lactulose: 15 mg of bisacodyl and 60 grams crystalline lactulose x 3 doses
- Total: Total of all reporting groups
Arm/Group | 90 Grams of Crystalline Lactulose | 135 Grams of Crystalline Lactulose | 180 Grams of Crystalline Lactulose | Total
Number analyzed (Participants) | 8 | 12 | 12 | 32
Age, Continuous [Mean (Standard Deviation); unit: years]
  Subject Age at Enrollment | 47.4 (6.2) | 57.0 (7.4) | 58.1 (8.7) | 55.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 9 | 21
  Male | 4 | 4 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 7 | 12 | 11 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 8 | 11 | 10 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Bisacodyl and Lactulose as a Preparation for Colonoscopy.
Description: Efficacy assessed by the physician's determination of the cleanliness of the colon using the Boston Bowel Preparation Scale (BBPS). 9 is the maximum score, representing an fully cleansed colon; 0 is the minimal score, representing a colon with no cleaning.
Time Frame: 10-14 hours post last consumption
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 90 Grams of Crystalline Lactulose | 135 Grams of Crystalline Lactulose | 180 Grams of Crystalline Lactulose
Number analyzed (Participants) | 7 | 12 | 12
units on a scale | 5.7 (2.8) | 7.4 (0.9) | 7.8 (0.8)

2. Secondary Outcome: Safety of Bisacodyl and Lactulose as a Bowel evacuant_AE Incidence
Description: Safety determined by the incidence of treatment emergent adverse events.
Time Frame: 1 day post last consumption
Measure: Number; unit: % of patients with adverse events
Arm/Group | 90 Grams of Crystalline Lactulose | 135 Grams of Crystalline Lactulose | 180 Grams of Crystalline Lactulose
Number analyzed (Participants) | 8 | 12 | 12
% of patients with adverse events | 25 | 33 | 50

3. Secondary Outcome: Safety of Bisacodyl and Lactulose as a Bowel evacuant_AE Severity
Description: Safety determined by the severity of treatment emergent adverse events.
Time Frame: 1 day post last consumption
Measure: Number; unit: Percentage of subjects
Arm/Group | 90 Grams of Crystalline Lactulose | 135 Grams of Crystalline Lactulose | 180 Grams of Crystalline Lactulose
Number analyzed (Participants) | 8 | 12 | 12
Percentage of subjects
  Mild | 0 | 25 | 50
  Moderate | 25 | 8 | 0
  Severe | 0 | 0 | 0

4. Secondary Outcome: Tolerability of and Preference for Bisacodyl and Lactulose as a Bowel Evacuant
Description: Tolerability assessed by a patient questionnaire. Overall tolerability as given by Visual Analog Scale (VAS): 100 represents maximally tolerable; 0 represents minimally tolerable
Time Frame: 1 day post last consumption
Measure: Mean (Standard Deviation); unit: units on a VAS scale
Arm/Group | 90 Grams of Crystalline Lactulose | 135 Grams of Crystalline Lactulose | 180 Grams of Crystalline Lactulose
Number analyzed (Participants) | 8 | 12 | 12
units on a VAS scale | 65.4 (27.6) | 68.5 (19.6) | 71.3 (18.4)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the first dose of study drug through the end of the observation period after the colonoscopy (Day 2).
Arm/Group | 90 Grams of Crystalline Lactulose | 135 Grams of Crystalline Lactulose | 180 Grams of Crystalline Lactulose
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/8 | 4/12 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 90 Grams of Crystalline Lactulose (N=8) | 135 Grams of Crystalline Lactulose (N=12) | 180 Grams of Crystalline Lactulose (N=12)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Procedural hypotension (Vascular disorders) | 0 (0) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No